CLINICAL TRIAL: NCT06766669
Title: Adapting Shaping Activities Into Mirror Therapy and Its Effects on Motor Dexterity, Motor Learning and Reaction Time in Healthy Individuals: A Case-Control Study
Brief Title: Adapting Shaping Activities Into Mirror Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MarmaraU-FTR; 1919B012210132 (Other Grant/Funding Number: TÜBİTAK, 2209-A- Research Project Support Programme for Undergraduate Students)
Record Dates: First submitted 2025-01-05; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-10

CONDITIONS: Healthy
Keywords: Mirror movement therapy; Motor activity; Motor skills; Reaction time
MeSH Terms: conditions — Motor Activity | interventions — Mirror Movement Therapy

STUDY DESIGN:
Intervention Model Description: Cross-Sectional, Case-Control Study Design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mirror Therapy Group (Experimental): In this group, Shaping Method activities are added to Mirror Therapy as a protocol and applied to participants.
  Interventions: Other: Shaping method activities combined with mirror therapy
- Control Group (No Intervention): The group that has no intervention and is asked to continue with their daily routines.

INTERVENTIONS:
Other: Shaping method activities combined with mirror therapy — This intervention involves the application of exercises consisting of shaping method activities accompanied by a mirror device. It is basically an intervention consisting of exercises that require manual dexterity.
  Arms: Mirror Therapy Group

SUMMARY:
The goal of this case-control study is to assess the impact of a novel method which adapts shaping activities into mirror therapy to improve dexterity, reaction time, and motor learning of the non-dominant hand in healthy individuals. The main question it aims to answer is:

Does the use of Shaping Method as a protocol in Mirror Therapy will have an enhancing effect on upper extremity motor skills, motor learning and reaction time in healthy individuals.

The objective of this study is to compare the intervention group, which will undergo shaping method activities in accordance with the protocol set out in Mirror Therapy, with the control group. This will enable an assessment of the impact of this approach on dexterity, reaction time and motor learning of the non-dominant hand in healthy individuals.

Participants in intervention group will:

* Use the Shaping Method activities with mirror therapy for 4 weeks.
* Come to the exercise lab 2 times a week for 4 weeks.
* Participate in assessment tests at the beginning and end of the intervention period.

Participants in control group will:

* Take assessment tests twice, four weeks apart.
* Maintain their daily routine for the duration of their participation in the study.

DETAILED DESCRIPTION:
In our study, 30 healthy adults were included in the intervention group and the same number of age- and gender-matched healthy adults were included in the control group.

The intervention group received 20-minute sessions, 2 days a week for 4 weeks. During the sessions, participants were seated with the non-dominant hand behind the mirror device and the dominant hand in front. The participants were instructed to perform the following exercises with their dominant hand for 10 repetitions in accordance with the Shaping Method: Clothespin attachment activity, Ring threading on rod, Connecting the dots, Putting pencils in the glass, Velcro board activity, Dipping fork in play dough activity, Placing the cubes in the box activity, Ball insertion into perforated plastic plate, The activity of touching colored paper placed between white papers, Geometric jigsaw activity. Participants were assessed with outcome measures before and at the end of the 4-week intervention period.

Participants in the control group received no intervention and were asked to continue their daily routines for 4 weeks. These participants were also assessed with outcome measures twice at 4-week intervals.

The SPSS 27.0 package program was used for statistical analysis. The normality of the distribution of quantitative variables was evaluated using the Shapiro-Wilk test. The demographic and clinical data were summarized as the mean ± standard deviation (SD) for the continuous variables and the number and percentage for the categorical variables. The initial measurements of the groups were compared using an independent samples t-test. A paired t-test was used to investigate intragroup differences between the pre- and post-tests. A one-way analysis of covariance (ANCOVA) was employed to determine the differences between the intervention and control groups, with baseline measurements serving as covariates. The differences between the groups were calculated based on the post-intervention assessment and the change from the pre-intervention values. The statistical significance was set to p< 0.05, and the effect sizes were interpreted as follows: ≤ 0.2, small; around 0.5, medium; ≥ 0.8, large.

ELIGIBILITY:
Inclusion Criteria:

* Between 18-30 years old
* Dominant limb is right

Exclusion Criteria:

* A history of orthopedic disease, neurological disease, and/or surgery of the upper extremities

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-07-26 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Roeder Manipulative Aptitude Test | From enrollment to the end of treatment at 4 weeks
  The Roeder Manipulative Aptitude Test, which involves the insertion of a rod, cap, washer, and nut-common field tools-into a perforated board, was employed to assess motor skills. The test is comprised of two phases, with a five-minute rest period between them. In the initial phase, which lasts three minutes, the subject is required to insert a rod and then a cap into the perforated sections with their non-dominant hand. The total number of rods and caps placed by the participant during this phase of the test is recorded as the unilateral score of the test. In the second stage of the test, which lasts 40 seconds, the participant places the nut and then the washer on the T-bar using both hands. At this juncture, the number of nuts and washers placed on the right and left sides is totaled and recorded as the bilateral score of the test. The sum of the unilateral and bilateral scores represents the total score of the test.

SECONDARY OUTCOMES:
Nelson Hand Reaction Time Test | From enrollment to the end of treatment at 4 weeks
  This Test was employed to assess the participants' reaction time. During the test, the participant was seated in a chair and extended the non-dominant hand, with the thumb positioned opposite the other fingers, 8-10 cm away from the table. The initial point of a 50-centimeter-long ruler was held between the participant's thumb and index fingers, and the participant was instructed to fixate the center of the ruler. The researcher grasped the upper portion of the ruler and instructed the participant to "Ready!" before releasing the ruler. The participant was instructed to close their fingers as soon as possible in an attempt to catch the falling ruler. The test was repeated five times, with the two lowest scores being excluded. The arithmetic mean of the remaining three scores was then calculated.
Finger Tapping Test | From enrollment to the end of treatment at 4 weeks
  The Finger Tapping Test was employed to assess motor learning. The test was created on the Psytoolkit online platform (https://www.psytoolkit.org). For the test, participants were seated in front of a laptop screen and instructed to place four fingers of their non-dominant hand (the fifth finger on the "1," the second finger on the "4") on the "1," "2," "3," and "4" keys on the keyboard. The subject was required to perform a series of keystrokes (4-1-3-2-4) that appeared on the screen for 10 seconds, as quickly and accurately as possible. The test was administered in 9 repetitions, with a 10-second rest interval between each repetition. The total number of sequences that the participant correctly keyed in 9 trials was recorded as the test score.

CONTACTS AND LOCATIONS:
Overall Officials: Burcu Ersöz Hüseyinsinoğlu, Associate Professor, Principal Investigator — Marmara University, Department of Physiotherapy and Rehabilitation; Özlem Doğan, Study Chair — Marmara University, Department of Physiotherapy and Rehabilitation; Alime Nur Kara, Study Chair — Marmara University, Department of Physiotherapy and Rehabilitation; Sergen Öztürk, MSc, Study Chair — Marmara University, Institute of Health Sciences
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jha RK, Thapa S, Kasti R, Nepal O. Influence of Body Mass Index, Handedness and Gender on Ruler Drop Method Reaction Time among Adults. J Nepal Health Res Counc. 2020 Apr 20;18(1):108-111. doi: 10.33314/jnhrc.v18i1.2545. PMID 32335603
- [Background] Aranha VP, Moitra M, Saxena S, Narkeesh K, Arumugam N, Samuel AJ. Motor cognitive processing speed estimation among the primary schoolchildren by deriving prediction formula: A cross-sectional study. J Neurosci Rural Pract. 2017 Jan-Mar;8(1):79-83. doi: 10.4103/0976-3147.193544. PMID 28149087
- [Background] Kesilmiş, İ., et al., Reaction Time in Target Shooting Sports: Perspective of Bocce and Archery. Eurasian Research in Sport Science, 2021. 6(2): p. 121-129.
- [Background] Çakıt, E., B. Durgun, and M. Cetik, Assessing the Relationship Between Hand Dimensions and Manual Dexterity Performance for Turkish Dental Students. Vol. 489. 2016. 469-479.
- [Background] Morris DM, Taub E, Mark VW. Constraint-induced movement therapy: characterizing the intervention protocol. Eura Medicophys. 2006 Sep;42(3):257-68. PMID 17039224
- See also: Related Info — https://clinicaltrials.gov/